CLINICAL TRIAL: NCT05054842
Title: Efficacy and Safety of Retagliptin Phosphate in Combination With Metformin in Type 2 Diabetic Subjects With Poor Metformin Glycemic Control: a Phase III Multicenter, Randomized, Double-blind, Placebo-controlled Design
Brief Title: Clinical Study of Retagliptin Phosphate Combined With Metformin in the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-SP2086-304
Record Dates: First submitted 2021-09-09; First posted 2021-09-23 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: SP2086 VS. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group A (Experimental)
  Interventions: Drug: Retagliptin phosphate tablets、metformin sustained-release tablets
- treatment group B (Placebo Comparator)
  Interventions: Drug: Retagliptin phosphate placebo tablets、metformin sustained-release tablets

INTERVENTIONS:
Drug: Retagliptin phosphate tablets、metformin sustained-release tablets — Retagliptin phosphate tablets 100mg+ metformin sustained-release tablets 1500mg or 2000mg based on prior medication
  Arms: treatment group A
Drug: Retagliptin phosphate placebo tablets、metformin sustained-release tablets — Retagliptin phosphate 100mg placebo tablets + metformin sustained-release tablets 1500mg or 2000mg based on prior medication
  Arms: treatment group B

SUMMARY:
Retagliptin phosphate tablet is a DPP IV inhibitor durg，study number is HR-SP2086-304. The primary purpose of the study is to evaluate the efficacy of the combination of Retagliptin phosphate and metformin compared with placebo and metformin in type 2 diabetes subjects with poor glycemic control treated with metformin for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent, understood the procedures and methods of the study, and was willing to complete the study strictly in accordance with the clinical trial protocol;
2. The screening age should be 18-75 years old (including both ends), male or female;
3. Diagnosed with type 2 diabetes, 7.5%≤HbA1c≤11%;
4. At least 8 weeks prior to screening, in addition to regular diet control and exercise, a steady dose of metformin ≥1500mg/d;
5. Fasting glucose ≤13.3mmol/L; 6、19.0 < BMI 35.0 kg/m2 or less.

Exclusion Criteria:

1. General situation:

   * 1) Known or suspected allergy to DPP4i drugs or investigational drug excipients;
   * 2) Pregnant or lactating women, fertile men or women were unwilling to use contraception during the study period;
2. History or evidence of any of the following diseases at the time of screening:

   * 1) Type 1 diabetes, single-gene mutation diabetes, diabetes due to pancreatic damage, or other secondary diabetes (e.g., diabetes due to Cushing's syndrome or acromegaly);
   * 2) Acute metabolic complications (such as ketoacidosis, lactic acidosis or hypertonic coma) occurred within 6 months prior to screening; Or have serious chronic complications of diabetes in the past (such as severe macrovascular or microvascular complications as judged by the investigator) and the investigator considers that they are not suitable to participate in this study;
   * 3) There is a history of severe hypoglycemia (such as drowsiness, disturbance of consciousness, delirium, or even coma caused by hypoglycemia, which requires the assistance of others for treatment), or repeated hypoglycemia (≥3 symptomatic hypoglycemia within a week, or blood glucose <3.0 mmol/L detected at least 3 times within a week);
   * 4) Patients with poorly controlled hypertension at screening were defined as systolic blood pressure (SBP) ≥160 mmHg and/or diastolic blood pressure (DBP) ≥100 mmHg;
   * 5) Had myocardial infarction, unstable angina, stroke (except lacunar infarction without attack symptoms) or transient ischemic attack, or had undergone coronary angioplasty, percutaneous coronary stent implantation or coronary artery bypass grafting within 6 months prior to screening; Or had congestive heart failure (NYHA grades III and IV), unstable or acute congestive heart failure, or persistent arrhythmias that the investigator determined significantly affected the subjects' safety within the 6 months prior to screening;
   * 6) History of acute and chronic pancreatitis, or risk factors that may lead to pancreatitis, such as history of symptomatic gallbladder, history of pancreatic injury, etc. (except cholecystectomy);
   * 7) A history of malignant tumor within 5 years prior to screening, excluding treated local basal cell carcinoma of the skin;
   * 8) have obvious diseases of the blood system (such as aplastic anemia, myelodysplastic syndrome, hemolytic anemia) or any diseases causing hemolysis or red blood cell instability (such as malaria);
   * 9) Clinically significant gastric emptying abnormalities (e.g., gastric outlet obstruction), severe chronic gastrointestinal diseases (e.g., active ulcers within 6 months prior to screening);
   * 10) There is a history of drug or alcohol abuse within 3 months prior to screening, which may affect the subject's compliance to participate in the test according to the investigator's judgment;
3. Received any of the following pharmacological or non-pharmacological treatments or procedures prior to screening:

   * 1) Any hypoglycemic drug treatment other than metformin within 2 months prior to screening, including Chinese herbal therapy for hypoglycemic purposes (except cumulative use ≤7 days);
   * 2) received systemic steroid hormone therapy (including intravenous and oral administration) and intraarticular administration for more than 7 days within 2 months prior to screening;
   * 3) Bariatric surgery or procedures (e.g. gastric banding surgery) within 12 months prior to screening, or use of weight-loss medications within 3 months prior to screening, or weight fluctuation ≥10% within 3 months prior to screening;
   * 4) Have received other gastrointestinal surgery that may lead to malabsorption before screening, or long-term use of drugs that directly affect gastrointestinal motility;
   * 5) Have received blood transfusion, blood donation or blood loss ≥400 mL within 3 months before screening;
   * 6) Participated in clinical trials of any drug or medical device within 3 months prior to screening (subject to entering into randomised procedures);
4. Any of the laboratory test indicators during screening meet the following standards (those who meet the criteria can be retested once within one week if there is a clear reason for retesting) :

   * 1) Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥3.0×ULN and/or total bilirubin ≥2.0×ULN;
   * 2) patients with renal function injury were defined as eGFR <60ml/min/1.73 m2 (calculated according to the simplified formula of dietary adjustment for renal disease (MDRD));
   * 3) Thyroid function test: abnormal thyroid stimulating hormone (TSH), serum free triiodothyronine (FT3), serum free thyroxine (FT4);
   * 4) Fasting triglyceride ≥5.64 mmol/L (500 mg/ dL);
   * 5) Blood amylase or lipase exceeded the upper limit of the normal range and was clinically significant as judged by researchers
5. Significant abnormal 12-lead electrocardiogram (ECG) results during screening, which the investigator considered might affect the safety of the subjects and are not suitable for this study;
6. Any other conditions (such as affecting the safety or efficacy evaluation of the subjects) that the investigator deemed inappropriate for the subjects to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c relative to baseline | After 16 weeks of treatment

SECONDARY OUTCOMES:
The proportion of subjects with HbA1c<6.5% and HbA1c< 7% after 16 weeks of treatment | up to 16 weeks of treatment
Changes in fasting plasma glucose relative to baseline | up to 16 weeks of treatment
Changes in 2h postprandial blood glucose relative to baseline | up to 16 weeks of treatment
Changes in body weight relative to baseline | up to 16 weeks of treatment
Percentage of subjects in each group who received remedial treatment | up to 16 weeks of treatment]
The incidence of adverse events of SP2086 | From Day 1 to Day 113
The incidence of Hypoglycemic event of SP2086 | From Day 1 to Day 113
Evaluate the concentrations of SP2086 in Type 2 diabetes | up to 16 weeks of treatment
Evaluate the concentration of the main metabolite of SP2086 in Type 2 diabetes | up to 16 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided